CLINICAL TRIAL: NCT06669091
Title: A Phase 1, Randomized, 2-way Crossover, Food-effect Study of Ecopipam Pharmacokinetics After Administration of the to Be Marketed Tablet in Healthy Subjects
Brief Title: Food-effect Study of Ecopipam Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EBS-101-HV-107
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Food-effect
MeSH Terms: interventions — ecopipam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dosed in fasted state (Other): Ecopipam will be taken in the morning in a fasted state
  Interventions: Drug: Ecopipam tablet
- Dosed in fed state (Other): Ecopipam will be taken in the morning after a standard high-fat breakfast
  Interventions: Drug: Ecopipam tablet

INTERVENTIONS:
Drug: Ecopipam tablet — A single ecopipam 89.6 mg tablet (equivalent to ecopipam HCl 100 mg)

SUMMARY:
Standard food-effect study to identify the effect of food on ecopipam pharmacokinetics after administration of a to-be-marketed ecopipam tablet in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects or female subjects of non-childbearing potential
* ≥18 and ≤55 years of age
* BMI >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
* Subjects must be healthy, as determined by the Investigator, based on medical history, physical examination, ECG, vital signs, and standard panel of blood and laboratory tests at Screening.
* Sexually active males must use a double barrier method of contraception during the study and for at least 90 days after the last dose of study drug.
* Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.

Exclusion Criteria:

* History of significant medical illness
* Clinically significant abnormalities on screening tests/exams
* History of or significant risk of committing suicide
* Donation of plasma within 1 month prior to dosing
* Donation or significant loss of blood within 8 weeks prior to the first dosing
* Major surgery within 3 months or minor surgery within 1 month prior to admission
* Use of prohibited prescription, over-the-counter medications or natural health products
* Use of tobacco or nicotine products within 1 month prior to Screening
* Significant alcohol consumption or history of abuse
* History of drug abuse within the previous 2 years, or a positive drug screen
* History of cannabinoid use within the previous 3 months
* Positive urine drug screen, urine cotinine test, or alcohol breath test
* History of allergy to study medications
* Recent participation in a clinical research study
* Prior exposure to ecopipam
* Not suitable for study in the opinion of the Principal Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Cmax of ecopipam after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of ecopipam after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC of ecopipam after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of ecopipam after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of ecopipam after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC of ecopipam after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of ecopipam after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis

SECONDARY OUTCOMES:
Cmax of EBS-101-40853 after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of EBS-101-40853 after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of EBS-101-40853 after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of EBS-101-40853 after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of EBS-101-40853 after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of EBS-101-40853 after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of EBS-101-40853 after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of EBS-101-40853 after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of ecopipam glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of ecopipam glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of ecopipam glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fed state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Tmax of EBS-101-40853 glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of ecopipam glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of ecopipam glucuronide after administration of an ecopipam tablet in the fasted state | Up to Day 13
  Up to 36 samples will be collected at the indicated time points for pharmacokinetic analysis
Safety and tolerability as demonstrated by concomitant medications | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Safety and tolerability as demonstrated by physical exams | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Safety and tolerability as demonstrated by AEs | Up to Day 20
  Subjects will be continually monitored for adverse events
Systolic blood pressure (SBP) and diastolic blood pressure (DBP) (mmHG) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Respiratory rate (breaths/minute) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Oral temperature (degrees Celsius) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Electrocardiogram (ECG) parameters: HR, PR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) (Milliseconds) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Values of white blood cell (WBC), neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets (1000/mm3) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Value of hematocrit (percent) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Value of hemoglobin (g/dL) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Red blood cell (RBC) count (M/mm3) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Values of bicarbonate, sodium, magnesium, potassium, chloride (mmol/L) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Values of urea, phosphorus, calcium, glucose, total cholesterol, HDL, LDL, triglycerides, uric acid, and total, direct and indirect bilirubin (mg/dL) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Values of albumin and total protein (g/dL) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Values of amylase, lipase, alanine aminotransferase (ALT), aspartate aminotransferase (AST),alkaline phosphatase (ALP), creatine phosphokinase (CPK), and creatinine (U/L) | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Value of urine pH | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Value of urine glucose | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Value of urine protein | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Value of urine blood | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints
Value of urine leukocyte esterase by dipstick | Up to Day 20
  Safety and tolerability measures will be recorded at the indicated timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Munschauer, MSc, MD, FAAN, Study Chair — Emalex Biosciences
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No